CLINICAL TRIAL: NCT06934473
Title: Effects of Endogenous GIP on Postprandial Blood Pressure in Healthy Individuals
Acronym: GA-25
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, lise wilki-kurtzhals, MD, PhD student, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: GA-25
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Bloodpressure
Keywords: Glucose-dependent insulinotropic polypeptide; GIP; GIP receptor antagonist; GIP(3-30)NH2
MeSH Terms: interventions — gastric inhibitory polypeptide (3-30)-amide; Sodium Chloride; gastric inhibitory polypeptide (1-42)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GIP(3-30)NH2 + mixed meal test (Experimental): Intravenous infusion of GIP(3-30)NH2 in a concentration of 1,000 pmol/kg/min + mixed meal test
  Interventions: Other: GIP(3-30)NH2 / study tool; Other: Saline (NaCl 0,9 %) (placebo)
- Saline + mixed meal test (Placebo Comparator): Intravenous infusion of saline 9 mg/ml added 0.5% human serum albumin + mixed meal test
  Interventions: Other: GIP(3-30)NH2 / study tool; Other: Saline (NaCl 0,9 %) (placebo)
- GIP(1-42) + water (Active Comparator): Intravenous infusion of GIP(1-42) in a concentration of 4,000 pmol/kg/min + intake of water
  Interventions: Other: GIP(1-42)
- Saline + water (Placebo Comparator): Intravenous infusion of saline 9 mg/ml added 0.5% human serum albumin + intake of water
  Interventions: Other: Saline (NaCl 0,9 %) (placebo); Other: GIP(1-42)

INTERVENTIONS:
Other: GIP(3-30)NH2 / study tool — Selective antagonist of the GIPR, GIP(3-30)NH2
  Arms: GIP(3-30)NH2 + mixed meal test; Saline + mixed meal test
Other: Saline (NaCl 0,9 %) (placebo) — Placebo (NaCl 0,9%)
  Arms: GIP(3-30)NH2 + mixed meal test; Saline + mixed meal test; Saline + water
Other: GIP(1-42) — Agonist of the GIPR, GIP(1-42)
  Arms: GIP(1-42) + water; Saline + water

SUMMARY:
The present study investigates the postprandial role of endogenous glucose-dependent insulinotropic polypeptide (GIP) on cardiovascular haemodynamics, hormone responses, and hypotensive symptoms during a tilt test.

DETAILED DESCRIPTION:
The study is an exploratory, randomised, placebo-controlled, double-blinded crossover study comprising four experimental days. Each experimental day consists of a mixed meal test or drinking water, a double-blinded continuous infusion of GIP(3-30)NH2 or placebo or GIP(1-42) or placebo, and three tilt tests. Sixteen healthy men and women will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-40 years
2. BMI between 18.5 and 29.9 kg/m2 (both included)
3. Informed consent

Exclusion Criteria:

1. Allergy or intolerance to ingredients included in the mixed meal
2. History of Orthostatic Hypotension (OH) or Postural Orthostatic Tachycardia Syndrome (POTS) or other autonomic dysfunction at the discretion of the investigators
3. Anaemia (haemoglobin below normal range <7.3 mmol/L for women and <8.3 mmol/L for men)
4. Kidney disease (estimated glomerular filtration rate (eGFR) <90 ml/min/1.73 m2) at screening
5. Known liver disease and/or elevated plasma alanine aminotransferase (ALT) > three times the upper limit of normal at screening
6. Treatment with antihypertensives
7. Treatment with GLP-1RA (Glucagon-like Peptide-1 Receptor Agonist)
8. Treatment with SNRI (Serotonin and Noradrenalin Reuptake Inhibitor) or treatment within two weeks before the first experimental day
9. Any ongoing medication that the investigator evaluates would interfere with trial participation
10. Any physical or psychological condition that the investigator evaluates would interfere with trial participation, including any acute or chronic illnesses
11. Any concomitant disease or treatment that, at the discretion of the investigators, might jeopardize the participant's safety during the trial
12. Alcohol/drug abuse as per discretion of the investigators
13. Pregnancy or breastfeeding
14. Participation in any other clinical trial during the study period
15. Mental incapacity or language barriers that preclude adequate understanding or cooperation or unwillingness to comply with trial requirements or pr discretion of the investigator

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Postprandial systolic blood pressure change (delta SBP) | From -35 to 50 minutes
  The mean difference between postprandial systolic blood pressure-change (delta SBP) during tilt test following infusion of GIP(3-30)NH2 compared to infusion of placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Copenhagen, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No